CLINICAL TRIAL: NCT02015130
Title: Individually Tailored Treatment of Type 2 Diabetes
Acronym: ITT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Odense University Hospital (Other)
Collaborators: Region of Southern Denmark (Other); Esbjerg Hospital - University Hospital of Southern Denmark (Other); General Practice Research Database (Other Government)
Responsible Party: Principal Investigator, Jacob Volmer Stidsen, MD, Odense University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Eudract2012-004883-23
Record Dates: First submitted 2013-12-03; First posted 2013-12-19 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Type 2 Diabetes; Hypertension
Keywords: Type 2 diabetes; hypertension; individual
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- individual treatment (Experimental): Individualized treatment
  Interventions: Other: Individual treatment
- control group (No Intervention): treatment according to current national guidelines

INTERVENTIONS:
Other: Individual treatment — See detailed description
  Other Names: mulitinterventional
  Arms: individual treatment

SUMMARY:
The prevalence of Type 2 diabetes (T2D) is rising rapidly worldwide. In Denmark approximately 8% of adults have T2D and more than 25.000 are diagnosed each year. This has vast consequences for society and the patient.

Standardized treatment aiming at normalizing blood glucose and hypertension comparable to healthy individuals, have been tested in large studies. The effect on cardiovascular disease and other complications have been modest at best and one study showed an increased mortality with intensive treatment. The standardized treatment often results in polypharmacy, which increases the risk of patients discontinuing treatment.

We propose a new approach to treatment of T2D, where the patients' individual characteristics are considered. The aetiology of the diabetes can be different, which warrants different treatment. Many patients have concomitant illness which can affect the way the patient is treated. A tight regulation of blood glucose can in some patient constitute a risk of adverse effects, especially hypoglycemia. In that sense individual targets for the treatment are important. Effective lifestyle treatment has importance for a successful outcome and we therefore offer an application that can help the patient and the physician organizing activity individually.

The objective of individual treatment is to choose the most effective medication. If a prescribed drug does not have the desired effect it should be replaced with a different drug. The overall goal is to reduce the number of substances and side-effects, but simultaneous improve treatment and reduce the incidence of cardiovascular and other diabetes-related complications. This will in turn result in improved quality of life and improved adherence to treatment.

The potential effect of individual tailored treatment of T2D is to improve the guidelines of treatment, not only to improve the patients' health, but also to reduce the socioeconomic consequences of the growing T2D prevalence

DETAILED DESCRIPTION:
The design is a prospective controlled open-label multicenter intervention study. General practitioners in region of southern Denmark are responsible for the treatment, while central visits for additional data sampling are located at Odense University hospital, Holbaek Hospital, Naestved Hospital, and hospital of south west Denmark, Esbjerg.

The inclusion phase will run for 2 years. The follow-up phase is 10 years from inclusion.

Registries will be employed in both the characterization of patients and in the sampling of end-points. Concomitant medication will be sampled from the National Prescription Database. Concomitant illness and identification of endpoints will be sampled from the Registry of Patients, Registry on Cause of Death, the Danish Registry on Regular Dialysis and transplantation, the Danish general practice database, The National Indicator project, Statistics Denmark, The National Indicator Project, The Danish Cancer Registry, the DD2-database and local databases.

Treatment The control group will be treated according to national guidelines. The intervention group will be treated according to individual assessment. Several approaches will be employed to achieve individualization.

* Identification of pathophysiological traits in order to chose the correct medication targeting hyperglycaemia. Identification of pathophysiological traits, through genetic testing, GAD antibodies and C-peptid level, will individualize the treatment of hyperglycaemia according to the following groups: MODY (maturity onset diabetes of the young), LADA (latent autoimmune diabetes of adults), steroid-induced diabetes, insulinopenic diabetes, secondary diabetes and patients with insulin resistance. Specific treatment algorithms will be applied in each group.
* Individualized targets for all patients with regard to hyperglycaemia. The target will be chosen on the basis of age, motivation, skills, risk of hypoglycaemic events, therapy resistance, initial hba1c and concomitant illness. As these factors change the target can be adjusted accordingly.
* Hemodynamic characterization by impedance cardiography will be used in order to individualize anti-hypertensive medication.
* Individualized targets for all patients with regard to hypertension. The target will be chosen on the basis of concomitant risk factors.

Further individualization will be achieved by discontinuing drugs which have not proven to be effective within a three-month period or have proven to have side-effects.

Treatment algorithms for the intervention group.

Hyperglycemia

* MODY (characterized by genetic test): Glimepiride or repaglinide for type 1 and 3. 1) diet, 2) basal insulin for type 2. Basal insulin for type 5
* LADA (GAD positive> 30UI/ml): basal bolus insulin-regime. Metformin if BMI > 25
* Secondary diabetes (HOMA-beta < 78.45 % AND history of pancreatitis or similar): basal bolus insulin regime
* Steroid induced diabetes: 1) meal time insulin 2) metformin 3) basal insulin if fasting blood glucose is above 7
* Insulinopenic type 2 diabetes (HOMA2-beta<78.45 % AND HOMA2-S>105.5%): 1) metformin 2) insulin, basal 3) meal time insulin
* Classical type 2 diabetes (HOMA2-beta<78.45% AND HOMA2-S<105.5%): 1) metformin 2) GLP-1 analogues* 3) basal insulin 4) meal time insulin.
* Hyperinsulinemic type 2 diabetes (HOMA2-beta>78.45% AND HOMA2-S<105.5%)

In patients with BMI>35 kg/m2 both gastric bypass and pharmacological treatment can be considered equally. In patients with BMI<35 kg/m2 only pharmacological treatment is an option:

1. In patients with BMI>35 kg/m2 gastric bypass should be considered according to the current national criteria and the preference of the patient.
2. 1) metformin 2) GLP-1 analogues* 3) Glitazones (pioglitazone is currently registered) 4) insulin, basal 5) meal time insulin If marked oedema develops in relation to institution of glitazones the treatment should be terminated. If patients have osteoporosis, glitazones should generally not be used.

If patients have heart failure glitazones should not be used.

*In cases were patients are reluctant to inject themselves or have economical objections, DD4-inhibitors can be chosen.

Premixed insulins can be used instead of basal insulin or instead of basal insulin+mealtime insulin whenever deemed relevant by the treating physician

Hypertension Hemodynamic characterization by impedance cardiography will be used in order to individualize anti-hypertensive medication. By impedance measures of vascular resistance, intravascular volemia and inotropy will be obtained.

All patients will be treated with ACE inhibitors. Secondary medication will in general be achieved by the following algorithm:

High vascular resistance:

1. Use ACE-inhibitor or add a calcium-channel blocker (CCB) to an existing ACE-inhibitor.
2. In case the resistance are increased by more than 100% and neither ACE-inhibitor or CCB is given, consecutive add both according to blood pressure. If hypervolemia is present address this before CCB is introduced.
3. If intravascular volume is normal and blood pressure is high after ACE-inhibitor; use CCB - also when resistance is normal

High intravascular volume:

1) Use hydrochlorthiazide 12.5mg combined with ACE inhibitor in one pill if possible. Else use bendroflumethiazide 2.5mg. If the patient is already receiving diuretics, spironolactone is used. Start with 25mg, maximum dose is 50mg. If kalium is above 4.3 or impaired kidney function is present start with 12.5mg. Control of kalium is paramount.

High inotropy

1) High inotropy might change with the institution of other drugs. Introduce CCB first and secondly thiazide if the patient is normovolemic. In reverse order if the patient is hypervolemic and with normal vascular resistance. Therefore high inotropy should only be treated with carvedilol if 1) the patient is receiving ACE inhibitor, thiazide and CCB and the impedance measure of high inotropy is made after ACE-inhibitor, thiazide and CCB is started.

Lifestyle A dietician will be employed to make written material regarding the diet. A Cookbook will be made available online, together with accompanying grocery lists. The diet will be done according to a composition of 20% protein, 40% fat and 40% carbohydrate to improve glycemic control. The extra percentage of fat, compared to current recommendations should come from polyunsaturated fat.

To facilitate exercise an accelerometer will be handed out and an individual goal of exercise will be set. A novel interface of the accelerometer will be used to monitor the exercise done and thereby enable the patient and the physician to evaluate the effort. Interval walking will be the general focus of the exercise guidance, if the patient does not have other individual exercise preferences. Individual goals of the exercise effort will be set and software will modify the goals according to current fitness.

Goal setting in the intervention group Treatment of hyperglycaemia should be made according to the following goals

* Optimal control of HbA1c < 6.5 % (48 mmol/mol)
* Acceptable control of hba1c < 7.5 % (58 mmol/mol)
* Free of symptoms, with the best possible Hb1ac within this restraint

The general practitioner is free to choose which goal is applicable, according to the above mentioned criteria. In patients with neuropathy or former cardiovascular disease extra vigilance should be taken if optimal control is chosen. If the patient develops a severe hypoglycaemic event, repeated measures of blood glucose below 4.0 mmol/l or is therapy resistant, the goal should be reassessed.

Treatment of hypertension should be made according to the following goals

1. BT < 135/85 in patients with microalbuminuria, increased creatinine or established cardiovascular disease
2. BT < 140/90 in patients without complications

First visit at primary physician In the control group this will be scheduled as deemed necessary by the physician In the intervention group this should be scheduled to be located after the baseline visit at the central hospital, in order to achieve collection of all relevant data for individualization.

Periodic visits at primary physician These are to take place every 3 month. At these visits treatment will be instituted according to the specified algorithms. If the goals are not met, intervals of 1 month are recommended in the intervention group.

Once a year the following will be collected for the study:

* Smoking habits, blood pressure, cholesterol levels, weight, HbA1c, Urine albumin-creatinine ratio, creatinine Visits for measurements of organ damage The initial visit will be scheduled within 4 weeks of the screening visit. Longitudinal measurements will be done after 2 and 4 years. The measurements will include
* ECG for assessment of ventricular hypertrophy
* Intima media thickness of the carotid artery along with assessment of plaque presence
* Measurement of calcification of the coronary arteries by heart CT (only year 0 and 4)
* Blood borne and urine markers of cardiovascular disease
* Automated office blood pressure (used to direct treatment)
* Ambulatory 24 hours blood pressure
* Questionnaire on quality of life, (at baseline: cardiovascular hereditary, former gestational diabetes or pancreatitis and prednisolon treatment within the last 3 month of debut)
* Thoracic impedans measurements
* Adverse events (side effects)
* medication
* Waist to hip ratio
* Fundus photo

These visits will be organized centrally. In a subset of patient echocardiography and pulse wave velocity will be performed.

Visits for measurements of thoracic impedans The measurement will be done after 0, 2, 4 (also after 1 year in the intervention group) years throughout the follow-up period and will be organized centrally.

Time schedule Oct 2013: Inclusion of patients Oct 2015: inclusion ends Oct 2019: analysis of surrogate markers of cardiovascular disease Oct 2025: sampling and analysis of endpoints

Cooperation between primary care and project coordinators Daily management and coordination will be handled by investigators at the 3 central hospitals. Data-sampling at central visits will be their responsibility. The central investigators will have an advisory role in the treatment of the patient. Initial pathophysiological characterization will be managed centrally and the results will be forwarded to the primary physician. The coordinating investigator will be responsible for gathering of data from registries.

The daily treatment of the patients will be managed by the primary physician according to the algorithms. Recruitment will also be done by the primary physician. Serious adverse events will be reported centrally by the GP.

TAP will be employed to do conduct the investigations at the central visits.

Concomitant illness and identification of endpoints will be sampled from the Registry of Patients, Registry on Cause of Death, the Danish Registry on Regular Dialysis and transplantation, The Danish general practice database, The National Indicator project, The Danish Cancer Registry, the DD2-database and local databases at time of analysis.

Concomitant illness will be established at the baseline visit through patient interview, aided by records from the Registry of Patients.

Endpoints will also be sampled real time as part of the sampling of SAEs.

Statistical considerations An incident rate of 2.5% per year of macro- and microvascular complications, of 1.5% for cancer and approximate 1% of over-all mortality is expected. Hypoglycaemic event rate is expected to be less than 0.4%. The expected incident rate of the composite endpoint is 5%, a power of 80% and a type I error of 0.05. A benefit of 20% with intervention is expected. Loss to follow-up: the database approach will limit this to a minimum. For a cumulated event rate of 5% during 10 years the estimated sample size is 1123 patients per group.

Ethical considerations The patient physical and mental integrity will be safeguarded. The participants will be protected by the law on personal data and the Danish health legislation act. The study will be conducted in compliance with the principles set forth in the declaration of Helsinki and the guidelines for god clinical practise (GCP). The Study will be conducted in compliance with this protocol as well as according to national legislation. The study will be approved by the regional committee on medical health ethics, the Danish data protection agency and the Danish Health and Medicines Authority. The study will be submitted at ClinicalTrial.gov.

ELIGIBILITY:
Inclusion Criteria:

1. Newly discovered diabetes patients clinically classified as T2D patients of both sex'
2. Participation in the DD2 cohort
3. Signed informed consent

Exclusion Criteria:

1. Patients with age under 18
2. Type 1 diabetes. If patients at baseline investigations have age<30 years AND C-peptid<300pmol/l AND GAD-ab titer> 20 IU/ml they are also considered as having type 1 diabetes.
3. Life expectancy below 2 years
4. Psychiatric or mental disease that affects the patients ability to give informed consent or participate adequately in the study
5. Ongoing abuse of alcohol or illicit drugs that affects the patients ability to give informed consent or participate adequately in the study
6. Participation in any other clinical trial
7. Pregnancy at time of inclusion or planned future pregnancy (A negative pregnancy test is mandatory before inclusion. In women who are sterile, infertile or is postmenopausal (12 month without menstruation) this test is omitted.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2246 (Estimated)
Dates: Start 2013-10; Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint: All cause mortality, non-fatal myocardial infarction, coronary revascularization, cardiac arrest with resuscitation, heart failure, non-fatal stroke, progression of nephropathy or retinopathy, severe hypoglycaemia and cancer | 10 year

SECONDARY OUTCOMES:
All cause mortality | 10 years
Socioeconomic cost | 10 years
Quality of life | 10 years

OTHER OUTCOMES:
Myocardial infarction, non-fatal | 10 years
Death from myocardial infarction | 10 years
Coronary revascularisation, CABG or PCI | 10 years
Heart failure: New, hospital admission due to acute deterioration (not related to new MI) or chronic regression in NYHA class | 10 years
Stroke or TCI, non-fatal | 10 years
Death from stroke | 10 years
Other revascularisation procedures | 10 years
Amputation due to macrovascular insufficiency | 10 years
Cardiac arrest with resuscitation | 10 years
Renal failure (defined by the need for chronic dialysis), development of macroalbuminuria, doubling of creatinine (only above 200) | 10 years
Proliferative retinopathy or macular oedema that require laser therapy, vitrectomy, diabetes related blindness (snellen visual acuity below 0.1) | 10 years
Severe hypoglycaemic events | 10 years
All-cause malignant cancer (not basocellular carcinoma) | 10 years
All cause hospitalization | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: jacob Stidsen, MD, Principal Investigator — Odense University Hospital; Henning Beck-Nielsen, Dr.med, MD, Study Chair — Odense University Hospital; Jeppe Gram, MD, Phd, Principal Investigator — Esbjerg Hospital - University Hospital of Southern Denmark; Jan Erik Henriksen, MD, Phd, Study Chair — Odense University Hospital; Jens Nielsen, PhD, Study Chair — Odense University Hospital
Locations (4):
- Denmark (4):
  - Hospital of south west Denmark, Esbjerg
  - Medicinsk afdeling.Holbæk Sygehus., Holbæk
  - Næstved Lægecenter, Næstved
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Norlen T, Olesen TB, Domazet SL, Nielsen JS, Brond JC, Olsen MH, Hojlund K, Stidsen JV. Physical activity and albuminuria in individuals recently diagnosed with type 2 diabetes. J Diabetes Complications. 2025 Aug;39(8):109065. doi: 10.1016/j.jdiacomp.2025.109065. Epub 2025 May 13. PMID 40398345
- [Derived] Domazet SL, Tarp J, Thomsen RW, Hojlund K, Stidsen JV, Brond JC, Grontved A, Nielsen JS. Accelerometer-derived physical activity and sedentary behaviors in individuals with newly diagnosed type 2 diabetes: A cross-sectional study from the Danish nationwide DD2 cohort. Front Sports Act Living. 2023 Jan 25;4:1089579. doi: 10.3389/fspor.2022.1089579. eCollection 2022. PMID 36761371
- [Derived] Stidsen JV, Nielsen JS, Henriksen JE, Friborg SG, Thomsen RW, Olesen TB, Olsen MH, Beck-Nielsen H. Protocol for the specialist supervised individualised multifactorial treatment of new clinically diagnosed type 2 diabetes in general practice (IDA): a prospective controlled multicentre open-label intervention study. BMJ Open. 2017 Dec 10;7(12):e017493. doi: 10.1136/bmjopen-2017-017493. PMID 29229652